CLINICAL TRIAL: NCT02026414
Title: Effects of PrimaVie and Exercise Training on Human Skeletal Muscle Adaptation
Brief Title: Effects of PrimaVie and Exercise Training on Human Skeletal Muscle (PrimaVie)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sanni Raju (Industry)
Collaborators: Ohio State University (Other)
Responsible Party: Sponsor-Investigator, Sanni Raju, CEO, Natreon, Inc.
Organization: Natreon, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 20131230
Record Dates: First submitted 2013-12-16; First posted 2014-01-03 (Estimated); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Obesity
Keywords: PrimaVie; Herbal Supplement; Muscle biopsy; Energy; Exercise; Human skeletal muscle adaptation; Muscle function
MeSH Terms: conditions — Obesity; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PrimaVie Exercise (Experimental): Subjects will take 250 mg of PrimaVie (herbal supplement manufactured by Natreon, Inc) twice a day for the first 8 weeks they are enrolled in the study. For the last 4 weeks of the study, subjects will take 250 mg of PrimaVie (herbal supplement manufactured by Natreon, Inc) supplement twice a day while also completing supervised exercise on a treadmill (70-75% of maximum Heart Rate for 20 mins, plus 5 minutes of warm up and 5 minutes of cool down exercises for a total of 30 minutes a day 3 days a week). Subjects will participate for a total of 12 weeks and come for three total visits. At each visit, subjects will have muscle biopsies taken from their thigh or calf as well as approximately 2 tablespoons of blood drawn.
  Interventions: Dietary Supplement: PrimaVie; Other: Exercise

INTERVENTIONS:
Dietary Supplement: PrimaVie — Subjects will take 250 mg of PrimaVie (herbal supplement manufactured by Natreon, Inc) twice a day for the first 8 weeks they are enrolled in the study. For the last 4 weeks of the study, subjects will take 250 mg of PrimaVie (herbal supplement manufactured by Natreon, Inc) supplement twice a day while also completing supervised exercise on a treadmill (70-75% of maximum Heart Rate for 20 mins, plus 5 minutes of warm up and 5 minutes of cool down exercises for a total of 30 minutes a day 3 days a week). Subjects will participate for a total of 12 weeks and come for three total visits. At each visit, subjects will have muscle biopsies taken from their thigh or calf as well as approximately 2 tablespoons of blood drawn.
  Other Names: purified and standardized shilajit extract
Other: Exercise

SUMMARY:
PrimaVie (Natreon Inc), is a a purified and standardized shilajit extract for nutraceutical use. Research indicates that PrimaVie® has targeted action for increasing energy, revitalization and anti-aging. Findings on a recent murine study revealed that PrimaVie (PV) significantly changed the expression of genes related to muscle function (unpublished data). Based on these facts, it was thought of interest to study the effect of PrimaVie and exercise training on human skeletal muscle adaptation.

The objective of the study is to determine effect of PrimaVie supplementation and combined PrimaVie supplementation and exercise on changes in muscle gene expression related to muscle function. Two hypothesizes have been made, oral supplementation of PrimaVie twice a day for 12 weeks will influence gene expression in the skeletal muscle of pre-obese to obese humans, oral supplementation of PV will act with treadmill exercise training to favorably impact skeletal muscle gene expression. The participants will have a total of 3 visits over 12 weeks. During each visit will include measurement of height, weight and vital signs, 2 tablespoons of blood will be draw from left or right arm, and muscle biopsies (using biopsy needle) will be collected under the use of local anesthetics. The blood and muscle biopsies will be used for all lab related procedure.

DETAILED DESCRIPTION:
Potential subjects will see an advertisement placed in locations around the Wexner Medical Center with RN (research nurse) listed as the main contact. After potential subjects contact the research nurse, he/she will use inclusion/exclusion criteria to determine potential eligibility. If the potential subject meets all inclusion/exclusion criteria, he/she will be scheduled for a primary visit at the Morehouse Medical Plaza or Davis Heart and Lung Research Institute. At this initial visit, the research nurse will meet the potential subject in a private room where the study will be fully explained in lay language, and informed consent will be obtained. Then, appropriate demographic, biometric and health/clinical information will be recorded on the data collection sheet, and 22.5 mL of blood will be obtained via venipuncture in the right/ left forearm. A muscle biopsy will also be collected by a trained physician. The blood and muscle biopsy will be used for all lab related study procedures. The subjects will be given an 8-week supply of the PrimaVie supplement with instructions, as well as a copy of the research protocol and informed consent form. If the supplements are mailed, they will also have instructions, as well as a copy of the research protocol and informed consent form mailed. The subject will be instructed to call the Research Nurse/ approved study personnel to let them know that they have received the supplements by mail and to go over any questions or concerns the subject may have as well as to schedule follow up visits. All follow up visits (T1, T2, T3a and T3b) will consist of a 22.5 mL blood draw, collection of muscle biopsy/biopsies and measurement of previously specified demographic, biometric and health/clinical variables.

For 4 weeks of exercise treadmill training (70-75% HRmax for 20 mins; 5 min warm up and 5 min cool down - total 30 mins a day; 3 days a week), the subjects will be doing supervised (study personnel) exercise routine (Treadmill) at study designated facilities( located on The Ohio State University campus).

Study Hypotheses:

* Hypothesis 1: That oral supplementation of PrimaVie twice a day for 12 weeks will influence gene expression in the skeletal muscle of sedentary pre-obese to obese humans
* Hypothesis 2: That oral supplementation of PrimaVie will synergistically act with treadmill exercise training to favorably impact skeletal muscle gene expression.

Aim: A non-randomized, longitudinal study to determine the effect of PrimaVie and exercise training on human skeletal muscle adaptation in 30 pre-obese to obese volunteers.

Participants: 40 volunteers will be recruited via study advertisement, and contact the research staff based on the study inclusion and exclusion criteria. At each visit the following will be recorded/collected:

* 22.5 mL of blood (approximately 2 tablespoons) (venipuncture)
* Muscle biopsy/biopsies (1 muscle biopsy per visit collected at T1 and T2, and 2 muscle biopsies are collected at T3)
* Age (years)
* Sex (M/F)
* Height (cm)
* Weight (lbs)
* BMI (Kg/m2)
* Blood pressure (mm/Hg)
* Pulse
* Body fat Percentage
* During the first visit (enrollment visit, T1), the following information will be recorded/collected as well:
* Tobacco use history
* Current alcohol use
* Current other drug use
* Current exercise regimen
* Date of first day of last menstrual period (for females only)
* Current Medications
* Allergies
* Nonmedical information, including: address (will be used to send PrimaVie supplement via mail, when applicable); telephone number, and email address

Participants will come for three visits:

* Visit 1 (T1) - Baseline (prior to the start of supplementation)
* Visit 2 (T2) - First 8 weeks of supplementation alone
* Visit 3 (T3) - Next 4 weeks of supplementation together with exercise (T3 consists of 2 sample collections: T3a (pre-exercise) after 12 weeks of supplementation together with 4 weeks of exercise - samples taken immediately before the final exercise routine (during Visit 3), and T3b (post exercise) after 12 weeks of supplementation together with 4 weeks of exercise immediately after the final exercise routine (during Visit 3)

Samples collected from participants:

* Peripheral blood: At all visits, 22.5 mL of peripheral venous blood will be collected.
* Muscle biopsies: biopsies will be collected from the Vastus lateralis or Gastrocnemius muscles. A biopsy will be collected by a board certified Physician after application of local anesthetic to the site of biopsy.

Study Supplement: PrimaVie (Natreon Inc), is a a purified and standardized shilajit extract for nutraceutical use. Research indicates that PrimaVie® has targeted action for increasing energy, revitalization and anti-aging. PrimaVie® also works at the cellular level, playing a direct role in the synthesis of ATP, a compound that supplies the body with energy, and healthy mitochondrial function. Findings on a recent murine study revealed that PrimaVie (PV) significantly changed the expression of genes related to muscle function (unpublished data). Based on these facts, it was thought of interest to study the effect of PrimaVie and exercise training on human skeletal muscle adaptation. Participants will take:

* 500 mg/day PrimaVie (Natreon Inc.) supplement, 250 twice a day for the first 8 weeks of the study( a 250 mg capsule in the morning with food and a 250 mg capsule in the evening with food)
* 500 mg/day PrimaVie (Natreon Inc) supplement, 250 mg twice a day for the next 4 weeks (a 250 mg capsule in the morning with food and a 250 mg capsule in the evening with food) of the study while including supervised exercise treadmill training, which includes:
* exercise supervised treadmill training (supervised treadmill training which include a 5 minute warm up; 70-75% HRmax for 20 minutes; and a 5 minute cool down - a total 30 minutes per day for 3 days per week)

ELIGIBILITY:
Inclusion Criteria:

* Patients 21-70 years of age
* BMI 25-34.9

Exclusion Criteria:

* BMI >35 OR < 25
* Individuals who are deemed unable to understand the procedures, risks and benefits of the study,( i.e. Informed consent) will be excluded
* Females who are pregnant as well as individuals who are therapeutically immuno-compromised will also be excluded in order to minimize the risk to such individuals (and fetus); to decrease statistical variability and to minimize potential of confounders.
* Candidates for inclusion into the study will not include individuals as defined in 45 CFR 46 Subparts B, C and D, nor from any other population which may be considered vulnerable. Pregnant women are excluded to minimize the risk to such individuals (and fetus); to decrease statistical variability and to minimize potential of confounders.
* History of MRSA (Methicillin-resistant Staphylococcus aureus)
* Current use of any of the following medications will result in exclusion:
* Steroids (Prednisone, etc.)
* Beta-Blockers
* Immunosuppressants
* Hydrochlorothiazide
* Statins (Crestor, Lipitor, etc.)
* Aspirin
* ACE Inhibitors
* Accutane (within the last 6 months)
* Muscle relaxants and stimulants

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-01; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Blood plasma assay | 12 Weeks
  Plasma creatine kinase (U/ml) myoglobin (ng/ml) troponin (ug/L) plasma glucose (mg/dl) lipid profiles (mg/dl) ATP levels (umol/L)
  Plasma creatine kinase, myoglobin, ATP and troponin will indicate muscle damage (these are "muscle damage markers").

SECONDARY OUTCOMES:
Muscle Biopsy Results | 12 Weeks
  Biopsies from the Vastus lateralis or Gastrocnemius muscles will be used for miRNA expression profiling (au) mRNA (delta Ct or fold change) protein determinations (fold change)

OTHER OUTCOMES:
BMI | 12 Weeks
  BMI (Kg/m2) Height, weight, age will be obtained and recorded at each visit for determination of BMI.

CONTACTS AND LOCATIONS:
Overall Officials: Gayle Gordillo, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center (Davis Heart and Lung Research Institute), Columbus, Ohio, United States

REFERENCES:
- [Derived] Das A, Datta S, Rhea B, Sinha M, Veeraragavan M, Gordillo G, Roy S. The Human Skeletal Muscle Transcriptome in Response to Oral Shilajit Supplementation. J Med Food. 2016 Jul;19(7):701-9. doi: 10.1089/jmf.2016.0010. PMID 27414521
- See also: Calculating Heart Rate Max — http://www.ntnu.edu/cerg/hrmax-info
- See also: OSU Wexner Medical Center Comprehensive Wound Center — http://medicalcenter.osu.edu/patientcare/healthcare_services/wound_care/Pages/index.aspx